CLINICAL TRIAL: NCT00849966
Title: Celecoxib for Pediatric Adenotonsillectomy: A Randomized Controlled Double Blinded Study
Brief Title: Celecoxib for Pediatric Adenotonsillectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Kimmo Murto, Deputy Academic Chief, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #09/10E
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Tonsillectomy; Adenotonsillectomy; Pain, Postoperative
Keywords: Celebrex; celecoxib; Cyclooxygenase Inhibitors; Anti-Inflammatory Agents Non-Steroidal; Adverse drug events; quality of life; Pain Postoperative; Tonsillectomy; Adenotonsillectomy; Otologic Surgical Procedures
MeSH Terms: conditions — Pain, Postoperative; Drug-Related Side Effects and Adverse Reactions | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Celebrex suspension
  Interventions: Drug: Celebrex suspension
- B (Placebo Comparator): Placebo
  Interventions: Drug: Celebrex suspension; Drug: Placebo

INTERVENTIONS:
Drug: Celebrex suspension — Patients will be randomized to receive celecoxib suspension 6 mg/kg one hour prior to their scheduled surgery. In addition the patient will receive seven weight-based doses of celecoxib (3 mg/kg) to be administered every 10-12 hours while the child is awake; the first dose being administered the evening of surgery.
  All participants will receive undergo and post surgery anesthetic treatment according to the usual standards of practice at CHEO.
  Other Names: celecoxib
Drug: Placebo — Patients will be randomized to receive placebo by mouth one hour prior to their scheduled surgery. In addition the patient will receive seven weight-based doses of the placebo to be administered every 10-12 hours while the child is awake; the first dose being administered the evening of surgery.
  All participants will receive undergo and post surgery anesthetic treatment according to the usual standards of practice at CHEO.
  Other Names: Ora-Blend
  Arms: B

SUMMARY:
The investigators' study will involve the administration of either placebo or celecoxib to children aged 2 to 18 years of age undergoing tonsillectomy and assessing pain relief, impact on quality of life and side effect profile.

DETAILED DESCRIPTION:
The study will consist of two arms, one placebo and the other celecoxib. To establish baseline data on the day of surgery the parents will be required to complete a validated parent report quality of life inventory, multi-dimension fatigue scale and pediatric pain questionnaire for the preceding week. Children/adolescents aged 8 to 18 years of age will be required to complete a child self-report of the same modules. Children undergoing adenotonsillectomy will receive either placebo or celecoxib by mouth one hour prior to their surgery. They will all receive preoperative acetaminophen. Premedication with midazolam will be at the discretion of the attending anesthesiologist. The patients will undergo a standardized anesthetic protocol including postoperative management of pain and nausea and vomiting. The patients, while under anesthesia, will have blood drawn to screen for occult liver and kidney disease, determine their CYP2C9 genotype and reserve for future gene chip micro array analysis.

Patients in both study arms will receive a second dose of celecoxib or placebo by mouth in the evening after surgery and then consecutively in the morning and evening for 72 hours. For seven days after the surgery the families will record once a day pain scores, document analgesic use and any side effects or adverse events. The families will be contacted by phone in the evening of the first three postoperative days to ensure that they understand and are completing the required documentation. On the seventh postoperative day the parents and children aged 8 to 18 years of age will be contacted by phone and instructed to complete the same two validated questionnaires concerning quality of life and level of fatigue completed on the day of surgery. Parents of children less than eight years of age will be responsible for completing these questionnaires based on observations of their children. On the 11th postoperative day the families will be contacted by e-mail or regular mail to complete a questionnaire asking about the extent of contact with the healthcare system, bleeding complications, recovery and overall satisfaction with their care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-18 years
* Tonsillectomy, or adenotonsillectomy
* No exclusion criteria

Exclusion Criteria:

* Age < 2yrs and >18yrs old
* BMI < 10th or > 95th percentile
* Serum creatinine (Cr) > 2 X UNL (upper normal limit)
* Abnormal liver function; namely alanine aminotransferase (ALT) > 1.5 X UNL, alkaline phosphatase (ALP) > 5X UNL, total bilirubin > 2 X UNL
* History of peptic ulcer disease.
* History of bleeding disorders
* History of severe asthma (requiring recent hospital admission or oral corticosteroid therapy)
* Allergy to celecoxib, sulfonamide compounds or NSAIDs
* Patients receiving CYP2C9 inhibitors fluconazole, amiodarone and oxandrolone
* Patients receiving CYP2C9 inducers rifampin and phenobarbital
* Extremes of body mass index (BMI) (age related below10th or above 90th percentile)
* Parents of any participants, irrespective of age, who are unable to read and understand instructions relayed in English or French
* Participant and/or parents of any participants, irrespective of age, who suffer from dementia, psychosis, significant developmental delay or other impairment that would prohibit the understanding and giving of informed consent or assent or the participation in self-care or toxicity reporting

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 282 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The investigators primary objective will be to determine the level of postoperative pain relief celecoxib provides for children within the first three days after undergoing tonsillectomy, or adenotonsillectomy | three days

SECONDARY OUTCOMES:
To measure the frequency of adverse events post surgery | For seven days immediately after the procedure
To quantify the impact of celecoxib on fatigue | Day 0 before the procedure and again on Day 7 afterwards
To quantify the impact of celecoxib on quality of life | Day 0 before the procedure and again on Day 7 afterwards
To quantify the impact of celecoxib on pain relief postsurgery | Day 0 before the procedure and every day until Day 7 afterwards
To identify polymorphisms of CYP2C9 genotypes and their impact on pain relief. | Sample taken during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Murto, MD, FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Murto K, Lamontagne C, McFaul C, MacCormick J, Ramakko KA, Aglipay M, Rosen D, Vaillancourt R. Celecoxib pharmacogenetics and pediatric adenotonsillectomy: a double-blinded randomized controlled study. Can J Anaesth. 2015 Jul;62(7):785-97. doi: 10.1007/s12630-015-0376-1. Epub 2015 Apr 7. PMID 25846344